CLINICAL TRIAL: NCT06561490
Title: Placental Thickness And Volume Nomogram In Normal Singleton Pregnancies Between 11th And 18th Week Gestational Age
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, hossam eldeen mostafa abdelkhalek, Resident in the Obstetrics and Gynecology Department Sohag university Hospital, Sohag University
Other Study IDs: Soh-Med-24-07-01MS
Record Dates: First submitted 2024-08-11; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Placental Volume

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- placental volume and thickness in normal singleton pregnancy
  Interventions: Radiation: sonographic assesment of placental thickness and volume

INTERVENTIONS:
Radiation: sonographic assesment of placental thickness and volume — sonographic assesment of placental thickness and volume

SUMMARY:
Measurement of placental thickness and volume has a great importance in predicting adverse outcome specially in combination with other markers.

In order to determine abnormalities in placental thickness and volume, we should have a normal range of values and this can be achieved by a nomogram

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies,11-18 weeks Reliable LMP Cases of ICSI with accurate date of transfer Cases of IUI with accurate date of IUI Cases of timed intercourse

Exclusion Criteria:

* Maternal Diseases Fetal anomalies Placenta previa, placental anomalies and poor visualization of the placenta Multiple pregnancies Unreliable gestational age

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Singleton pregnancies,11-18 weeks Reliable LMP Cases of ICSI with accurate date of transfer Cases of IUI with accurate date of IUI Cases of timed intercourse
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
placental thickness | 6 months
  placental thickness in normal singleton pregnancy between 11th and 18 th week gestational age
placental volume | 6 months
  placental volume in normal singleton pregnancy between 11th and 18 th week gestational age

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karthikeyan T, Subramaniam RK, Johnson W, Prabhu K. Placental thickness & its correlation to gestational age & foetal growth parameters- a cross sectional ultrasonographic study. J Clin Diagn Res. 2012 Dec;6(10):1732-5. doi: 10.7860/JCDR/2012/4867.2652. Epub 2012 Dec 15. PMID 23373039
- [Background] Wolfson RN, Zador IE, Halvorsen P, Andrews B, Sokol RJ. Biparietal diameter in premature rupture of membranes: errors in estimating gestational age. J Clin Ultrasound. 1983 Sep;11(7):371-4. doi: 10.1002/jcu.1870110705. PMID 6415121